CLINICAL TRIAL: NCT02981615
Title: A Phase 3, Multicenter, Randomized, Double Blind, Placebo Controlled Study to Assess the Safety and Efficacy of Antibacterial Prophylaxis for Prevention of Infections in Azacitidine Treated Myelodysplastic Syndrome Patients.
Brief Title: Phase 3 Multicenter Randomized Double Blind Placebo Controlled Study With Antibacterial Prophylaxis in Azacitidine Treated MDS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Drorit Merkel, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1680-14-SMC
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Prevention
MeSH Terms: interventions — Levofloxacin; Ofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental): Subjects allocated to the treatment arm of the study will be administrated Levofloxacin 500mg/d given p.o. once a day, starting on day 10 from beginning of each cycle until day 28 on an ambulatory basis. Levofloxacin will be continued in the first 4 Azacytidine cycles.
  Interventions: Drug: Levofloxacin
- placebo (Placebo Comparator): Subject allocated to the placebo arm will be treated with placebo once a day, starting on day 10 from beginning until day 28 of each of the first 4 cycles.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Levofloxacin — one tablet (500mg) a day, from day 10 to day 28 in every cycle of the 4 first cycles
  Other Names: levo, tavanic
  Arms: treatment arm
Drug: Placebo Oral Tablet — one tablet a day, from day 10 to day 28 in every cycle of the 4 first cycles
  Arms: placebo

SUMMARY:
Infections are a major and prevalent life-threatening complication among patients with myelodysplastic syndrome (MDS). Currently, the role of prophylactic antibacterial agents after chemotherapy in MDS patients remains controversial and there are no clinical guidelines for infection prophylaxis in this clinical setting. We will conduct a prospective study to evaluate the potential benefit of prophylactic antibacterial (Levofloxacin) on the rate of febrile episodes/infections in Azacytidine treated MDS patients.

DETAILED DESCRIPTION:
This is a national, multicenter, phase III, randomized, parallel arms, double blind, placebo controlled clinical trial to evaluate the efficacy and safety of antibacterial prophylaxis - Levofloxacin 500mg/d given p.o.in newly diagnosed MDS patients who are more than 18 years of age and fulfil an indication for Azacytidine treatment. Patients will be treated for up to 4 cycles of Levofloxacin, or placebo. Subjects allocated to the treatment arm of the study will be administrated Levofloxacin 500mg/d given p.o. once a day, starting on day 10 from beginning of each cycle until day 28. Subject allocated to the placebo arm will be treated with placebo once a day, starting on day 10 from beginning of each cycle until day 28. Levofloxacin and placebo treatment will be continued in the first 4 Azacytidine cycles. This study consists of 3 periods for each study subject: pre-treatment period, treatment period and follow up period. Expected duration of subject participation is 6 months Pre-treatment period: Assessments: MDS evaluation by bone marrow examination including cytogenetics/ FISH must be performed within half a year of the first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at the time of signing the informed consent document.
2. Have a documented diagnosis of primary or secondary MDS according to WHO 2008 classification (appendix I), fulfilling an indication for Azacytidine treatment.
3. Females of childbearing potential (FCBP) may participate, providing they meet the following conditions: Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study, and for 3 months following the last dose of study drug; and have a negative serum or urine pregnancy test (investigator's discretion; sensitivity at least 25 mIU/mL) at screening; and have a negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting study therapy in the treatment phase (note that the screening serum pregnancy test can be used as the test prior to starting study therapy in treatment phase if it is performed within the 72-hour time frame).
4. Male subjects with a female partner of childbearing potential must agree to the use of at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last dose of study drug.
5. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
6. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

Prior treatment with any of the following:

1.1. Azacitidine (any formulation), decitabine or other hypomethylating agent 1.2. Lenalidomide 2. Prior allogeneic or autologous stem cell transplant 3. Use of hydroxyurea within 7 days prior to randomization. 4. Diagnosis of AML (i.e. >30% blasts in bone marrow). 5. Ongoing adverse events from previous treatment, regardless of the time period. 6. Systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment) 7. Known Human Immunodeficiency Virus (HIV) 8. Known or suspected hypersensitivity to azacitidine or mannitol. 9. Known or suspected hypersensitivity to Levofloxacin. 10. Pregnant or lactating females. 11. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study. 12. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study. 13. Participation to an investigational drug trial in the last month before randomization.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Febrile episodes (fever >38.0c) rate. | from study entry to 6 months later

SECONDARY OUTCOMES:
Time to first febrile episode | from study entry to 6 months later
Clinically-documented (CDI) or microbiologically documented infections rate (MDI) | from study entry to 6 months later
  Clinically-documented (CDI) or microbiologically documented infections (MDI) other than bacteremia, defined as sepsis inflammatory response syndrome (SIRS) associated with local inflammation (e.g. pneumonia, UTI, abdominal infection) with or without microbiological documentation from the site of infection, excluding episodes accompanied by bacteremia. Virologically documented infections will not be included as MDIs
Bacteremia rate | from study entry to 6 months later
  Bacteremia, defined SIRS accompanied by growth of a bloodstream isolate in one or more blood culture. Growth of typical skin commensals (coagulase-negative Staphylococci, diphtheroids) will require growth from at least two separate sets of blood cultures.
Invasive fungal infections rate, as defined by the EORTC/MSG consensus group | from study entry to 6 months later
Number of participants use of antibacterial therapy other than levofloxain prophylaxis. | from study entry to 6 months later
Episodes of diarrhea rate | from study entry to 6 months later
C. difficile infection rate | from study entry to 6 months later
MDIs or bacteremia caused by quinolone-resistant bacteria rate | from study entry to 6 months later
Hospitalization for infection rate. | from study entry to 6 months later
Six months overall survival rate. | from study entry to 6 months later
QOL as measured by the FACT An questioner. | from study entry to 6 months later

OTHER OUTCOMES:
Correlation between serum ferritin level (> 1000ng/ml) as a predictor of the infection rate | from study entry to 4months later
Correlation between serum ferritin level (> 1000ng/ml) as a predictor of mortality rate | from study entry to 6 months later
Correlation of antibiotic prophylaxis use versus placebo on the rate of infections | from study entry to 6 months later
Correlation of antibiotic prophylaxis use versus placebo on the mortality rate | from study entry to 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Drorit G Merkel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chim Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No